CLINICAL TRIAL: NCT03314623
Title: Immediate Mobilization After Plate Osteosynthesis of Proximal Tibial Fractures - A Cohort Study
Acronym: IMOP
Status: Completed | Type: Observational
Sponsor: Slagelse Hospital (Other)
Responsible Party: Principal Investigator, Eske Brand, Doctor, Slagelse Hospital
Other Study IDs: 59459
Record Dates: First submitted 2017-10-09; First posted 2017-10-19 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Surgery--Complications; Tibia Fracture; Early Ambulation
MeSH Terms: conditions — Tibial Fractures | interventions — Weight-Bearing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Weight bearing as tolerated — If fracture is deemed stable the subjects will be allowed to weight bear immediately after surgery.

SUMMARY:
The purpose of this study is to investigate if immediate mobilization with weight bearing as tolerated following surgery with plates and screws after a fracture of the shinbone near the knee is possible without increased risk.

The investigators hypothesize immediate weight bearing as tolerated following surgery with plates and screws of the above mentioned fracture, in cases deemed stable by the surgeon, will not lead to any loss of reduction.

DETAILED DESCRIPTION:
The purpose of this study is to investigate immediate mobilization with weight bearing as tolerated following plate osteosynthesis after a proximal tibial plateau fracture is possible without increased risk of loss of reduction and/or failure of the osteosynthesis. Subsequently, this may lead to earlier recovery and less risk of thromboembolic complications.

The investigators hypothesize immediate weight bearing as tolerated (WBAT) following plate osteosynthesis after a proximal tibial plateau fracture, in cases deemed stable by the surgeon, will not lead to any loss of reduction.

Exposure will be defined as surgery with one or two angular stable plates (closed reduction, internal fixation) after a proximal tibial fracture. Patients will be allowed immediate weight bearing as tolerated in cases where the osteosynthesis is deemed stable. This represents the current practice at Slagelse Hospital. Typical, all lateral tibia plateau fractures (AO fracture classification 41B1-3) osteosynthesized will be allowed immediate WBAT after surgery. Other tibia plateau fractures will be allowed immediate WBAT if the osteosynthesis is deemed stable by the surgeon perioperatively.

Fractures are treated with one or several locking plates, and if needed after reduction of the tibial plateau, an impacted allogenic bone graft is used. The bone graft is applied through a cortical window osteotomy distal to the fracture.

Follow up will be performed at 2 weeks, 6 weeks, 3 months, 6 months and 1 year by any of the authors or a consultant in orthopedics. Follow up will be performed at the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized and osteosynthesized with one or several locking plates because of a proximal tibial fracture

Exclusion Criteria:

* Non-ambulatory patients,
* Patients diagnosed with dementia and
* Patients residing to another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient hospitalized at Slagelse hospital with proximal tibial fracture needing surgery with plates and screws residing in Slagelse hospital uptake area
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Loss of reduction | Day 0 to one year after surgery.
  Loss of reduction/fracture collapse after ambulation measured by x ray

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | Day 0 to one year after surgery.
  KOOS is a self-reported questionnaire comprising five subscales: pain, other symptoms, activities in daily living (ADL), function in sport and recreation and knee-related quality of life (QOL). The previous week is taken into consideration when patients are answering the questions. Standardized answer options are given (5 boxes on a Likert scale) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Return to Work | Day 0 to one year after surgery.
  If the subject hasnt worked prior to surgery, normal activity will be measured instead.
Length of Hospital Stay | Day 0 to one year after surgery.
Euroqol 5 Dimension (EQ-5D) | Day 0 to one year after surgery.
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The University of California at Los Angeles (UCLA) Activity Score | Day 0 to one year after surgery.
  A Danish version of the UCLA activity score will be used to assess the activity level before and after they have undergone surgery. The patients will answer the questionnaire preoperative and at the appointments in the outpatient clinic. The UCLA activity score ranges from 1-10 (not active-highly active) and the patient has to choose one out of the ten options based on their activity level for the past four weeks.
Radiographic Osteoarthritis | Day 0 to one year after surgery.
  Kellgren and Lawrence score
Status of reoperation | Day 0 to one year after surgery.
Performance Measures | Day 0 to one year after surgery.
  Knee range of motion
Status of surgery for acute compartment syndrome | Day 0 to 2 weeks after
Wound rupture | Day 0 to 6 weeks after
  Wound rupture needing suturing based on the evaluation by the investigators or a senior consultant
Infection | Day 0 to one year after surgery.
  Infection needing antibiotics, based on clinical findings combined with blodsamples measuring CRP and leucocytes.
Symptomatic deep venous thrombosis (DVT) | Day 0 to 6 weeks after
  Symptomatic DVT will be verified/disproved by ultrasound of the lower leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Slagelse Sygehus, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: Undecided